CLINICAL TRIAL: NCT05237440
Title: Childhood Traumas in Obese Women: Association With Deregulation of the Glucocorticoid Axis and Inflammatory State.
Acronym: OBEVIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 87RI21_0055 (OBEVIE)
Record Dates: First submitted 2022-01-07; First posted 2022-02-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Obesity
Keywords: obesity; childhood trauma; hypothalamic-pituitary-adrenal axis; inflammation; metabolic syndrome
MeSH Terms: conditions — Obesity; Inflammation; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other): Metabolic, hormonal and psychometric evaluations will be carried out during or after hospitalization inflammatory parameters, hormonal, capillary, saliva and urine assays will also be carried out
  Interventions: Biological: Biological dosage

INTERVENTIONS:
Biological: Biological dosage — Metabolic, hormonal and psychometric evaluations will be carried out during inclusion inflammatory parameters, hormonal, capillary, saliva and urine assays will also be carried out at inclusion

SUMMARY:
We postulate that childhood traumas are associated with deregulation of the glucocorticoid axis and the inflammatory system in obese women. The main objective of the study is to compare the salivary cortisol awaking response in obese women according to the presence of childhood trauma (assessed using the Childhood Trauma Questionnaire, CTQ).

DETAILED DESCRIPTION:
Obesity is an epidemic disease whose onset and development factors go beyond the simple energy balance. Current management strategies are often failing. It is therefore important to identify the underlying determinants of weight gain. The association of obesity in adulthood with trauma in childhood is now well established. However, the biological factors that account for this association are imperfectly known. The measurement of cortisol seems to be the most relevant biological marker of the link between obesity and life events. The majority of studies show that obesity is associated with increased exposure to glucocorticoids. However, some authors have recently reported that these measures are impacted by significant inter-individual variability which could be explained by differences in life events and especially in their perception. In addition, the autonomic nervous system with the secretion of catecholamines by the adrenal leads to the release of pro-inflammatory cytokines, resulting in a low grade inflammation.

The existence of childhood traumas and the association with other psychopathological disorders will be assessed using psychometric scales validated in French. The corticotropic axis will be evaluated by measuring cortisol in different matrices (saliva, urine, hair). The inflammatory state will be studied thanks to the determination of pro-inflammatory cytokines level in blood and immunophenotyping of myeloid-derived suppressor cells.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years female BMI≥30kg/m2

Exclusion Criteria:

1. History of bariatric surgery
2. Any condition or pathology that may influence the corticotropic axis or that may modify the excretion or dosage of cortisol:

   * pregnancy, breastfeeding
   * hepatocellular insufficiency,
   * severe heart failure,
   * mild/moderate acute heart failure,
   * any psychological disorder not stabilised for at least one year
   * alcohol or drug dependence, not weaned for at least one year
   * neoplasm under treatment
3. Current infectious disease or a history of autoimmune disease (except autoimmune hypothyroidism), inflammatory disease and/or neurodegenerative disease
4. Presence of an adrenal adenoma or any known or suspected clinical adrenal or corticotropic disorder
5. Subjects with a positive diagnosis of hypercorticism or suspected hypercorticism will also be excluded: 8-hour plasma cortisol after Dexamethasone suppression test (DST) (1 mg dexamethasone taken orally at midnight the previous day) greater than 1.8 microg/100 ml (50 nmol/l)
6. antidepressant and neuroleptic treatment, benzodiazepine treatment
7. treatment(s) likely to modify the exploration of the corticotropic axis: systemic or local corticosteroid therapy or glucocorticoid infiltration for less than 6 months
8. current use of anti-inflammatory drugs or antibiotics
9. Shift worker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-05-13 (Estimated); Study Completion 2024-05-13 (Estimated)

PRIMARY OUTCOMES:
Measurement of salivary cortisol awakening response (CAR) | Day 0
  Two salivary sampling at Day 0. The CAR is defined as the difference between the value of salivary cortisol collected 30 minutes after waking up and that on waking

SECONDARY OUTCOMES:
Comparison of the amount of urinary free cortisol | Day 21
  Comparison of the amount of urinary free cortisol in obese women according to the presence of childhood trauma (assessed using CTQs)
Comparison of the amount of urinary free cortisol metabolites | Day 21
  Comparison of the amount of urinary free cortisol metabolites in obese women according to the presence of childhood trauma (assessed using CTQs)
Comparison of the amount of salivary cortisone | Day 21
  Comparison of the amount of salivary cortisone in obese women according to the presence of childhood trauma (assessed using CTQs)
Comparison of the amount of hair cortisol/cortisone | Day 21
  Comparison of the amount of hair cortisol/cortisone in obese women according to the presence of childhood trauma (assessed using CTQs)
comparison of the proportions of current anxiety/depression | Day 0
  comparison of the proportions of current anxiety/depression with Hospital Anxiety and Depression Scale according to the presence of childhood trauma (assessed using CTQs). This scale includes14 items rated from 0 to 3. Questions are separated in two categories, 7 for anxiety and 7 for depression. thus allowing 2 scores to be obtained with a maximum of 21 for each.
comparison of the proportions of current post-traumatic stress disorder (PTSD) | Day 0
  comparison of the proportions of current post-traumatic stress disorder with PCL-5 scale according to the presence of childhood trauma (assessed using CTQs)
comparison of the proportion of current eating disorders | Day 0
  comparison of the proportion of current eating disorders with Dutch Eating Behavior Questionnaire according to the presence of childhood trauma (assessed using CTQs)
Dosage of several parameters of inflammation (CRP, IL-1beta, IFN-alpha2, IFN-gamma, TNF-alpha, CCL2 (MCP-1), IL-6, CXCL8 (IL-8), IL-10, IL-12p70, IL-17A, IL-18, IL-23, l'IL-33, T lymphocytes and Myeloid-Derived Suppressor Cells immunophenotyping) | Day 21
  Comparison of the parameters of inflammation in obese women according to the presence of childhood trauma (assessed using CTQ)
comparison of body composition | Day -7
  comparison of body composition in obese women by biphotonic absorptiometry according to the presence of childhood trauma (assessed using CTQ)
Comparison of the choice of treatment modality | Day 21
  Comparison of the choice of treatment modality (medical or surgical) according to the presence of childhood trauma (assessed using CTQ)

CONTACTS AND LOCATIONS:
Locations (1):
- LimogesUniversity Hospital, Limoges, France